CLINICAL TRIAL: NCT05037279
Title: A Multicenter, Randomized, Double-blind, Controlled Phase III Non-inferiority Study Assessing Efficacy and Safety of VERITY-BCG in Management of Intermediate and High-risk Non-muscle Invasive Bladder Cancer (NMIBC) in BCG-naïve Patients.
Brief Title: Evaluating Safety and Efficacy of Verity-BCG in BCG-naïve Patients with Intermediate and High-risk Non-muscle Invasive Bladder (NMIBC)
Acronym: EVER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Verity Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRT-BCG-01
Record Dates: First submitted 2021-07-28; First posted 2021-09-08 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer; Bladder Cancer Recurrent; Neoplasm Recurrence; Urothelial Carcinoma Bladder; Urothelial Carcinoma Recurrent; Non-Invasive Bladder Urothelial Carcinoma
Keywords: Interventional; Non-inferiority study
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verity-BCG (Experimental): * Bacillus Calmette-Guérin (BCG): Strain Russian BCG-I
  * Freeze-dried powder for bladder instillation
  Interventions: Drug: Bacillus Calmette-Guerin: Strain Russian BCG-I
- OncoTICE (Active Comparator): * Standard of Care
  * Bacillus Calmette-Guérin (BCG): Strain TICE
  * Freeze-dried powder for bladder instillation
  Interventions: Drug: Bacillus Calmette-Guerin: Strain TICE

INTERVENTIONS:
Drug: Bacillus Calmette-Guerin: Strain Russian BCG-I — * Induction: 80 mg weekly for 6 weeks.
  * Maintenance for intermediate AUA risk patients will be for 3 weeks at 3, 6, and 12 months.
  * Maintenance for high AUA risk patients will be for 3 weeks at 3, 6, 12, 18, 24, 30 and 36 months.
  Other Names: Verity-BCG
  Arms: Verity-BCG
Drug: Bacillus Calmette-Guerin: Strain TICE — * Induction: 50 mg weekly for 6 weeks.
  * Maintenance for intermediate AUA risk patients will be for 3 weeks at 3, 6, and 12 months.
  * Maintenance for high AUA risk patients will be for 3 weeks at 3, 6, 12, 18, 24, 30 and 36 months.
  Other Names: OncoTICE
  Arms: OncoTICE

SUMMARY:
The aim of this study is to evaluate the effect of Verity-BCG in patients with intermediate and high-risk non-muscle-invasive bladder cancer (NMIBC) and to compare our findings to the standard of care BCG formulation, OncoTICE (BCG) in order to examine our hypothesis that Verity-BCG is at least non-inferior to OncoTICE in achieving 24-month Recurrence Free Survival in NMIBC patients who are at high risk of recurrence and have never been treated with intradermal or intravesical BCG before, with the exception of tuberculosis vaccination in childhood.

DETAILED DESCRIPTION:
This study is a randomized, active control, double-blind clinical trial aimed at demonstrating non - inferiority of VERITY-BCG to OncoTICE, the current standard of care, with respect to two-year Recurrence Free Survival (RFS) rates in NMIBC BCG - naïve patients that are at high risk for recurrence (defined as >50%).

• Recurrence will be defined as the reappearance of any of the NMIBC tumors as confirmed by cystoscopic biopsy or TURBT.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years and older
* Low or high-grade NMIBC as defined by 2004 World Health Organization (WHO)/International Society of Urological Pathology (ISUP) classification and Grade 2 or 3 in the 1973 classification, diagnosed within 60 days of registration.
* Pathologically confirmed and completely resected stage Ta or T1 urothelial cell carcinoma, with or without associated carcinoma in situ (CIS), diagnosed within 60 days of registration.

  1. Patients with T1 disease must have imaging demonstrating no evidence of metastatic disease (based on MRI or CT scan) within 90 days of registration, to confirm stage T1N0M0 disease.
  2. For patients with stage T1 disease, repeat TURBT must be performed as per standard of care/CUA guidelines.
* Patients may have intermediate or high recurrence risk disease, as indicated by the probability of 2-year recurrence of ≥ 50% based on the EORTC Bladder Cancer risk calculator.
* ECOG performance status of 0-2
* Adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 unless data exists supporting safe use of BCG at lower kidney function values, no lower than 30 mL/min/1.73 m2
* For women of childbearing potential involved in any sexual intercourse that could lead to pregnancy: Negative pregnancy test and willingness to use contraceptive (consistent with local regulations) during 120 days after the last dose of the study treatment. Note: The use of contraceptive methods does not apply to subjects who are abstinent for at least 4 weeks before Day 1 and will continue to be abstinent from penile-vaginal intercourse 120 days after last dose of study drug treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.
* Note: A woman of non-childbearing potential is defined as follows:

  * Has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy);
  * Has had a cessation of menses for at least 12 months without an alternative medical cause, and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (refer to laboratory reference ranges for confirmatory levels).
* Male patients with female partner of childbearing potential must agree to be abstinent or practice an effective method of contraception.

Male patients must agree to refrain from donating sperm during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

* Presence of urothelial carcinoma involving the upper urinary tract or prostatic urethra documented by radiological imaging or biopsy, performed within 12 months of the start of treatment. Should the imaging or biopsy be performed outside the window it will be up to the physicians' discretion to re-scan/biopsy. This is considered T4 disease.
* CIS only disease.
* Pure squamous cell carcinoma or adenocarcinoma.
* Presence of micropapillary components.
* Other prior non-bladder malignancy, except for the following:

  * adequately treated basal cell or squamous cell skin cancer.
  * in situ cervical cancer.
  * adequately treated stage I or II cancer currently in complete remission, or any other cancer from which the patient has been disease free for five years.
  * patients with localized prostate cancer who are being followed by an active surveillance program are also eligible.
* Prior intravesical BCG or intradermal BCG, with the exception of tuberculosis vaccination in childhood.
* Chronic administration of steroids (>10 mg prednisone) at the time of randomization.
* Current or planned concomitant biologic therapy, radiation therapy, hormonal therapy, chemotherapy, surgery, or other cancer therapy while on study.
* Prior chemoradiation treatment (trimodal therapy or "TMT") for bladder cancer.
* Currently being treated or scheduled to have treatment with any systemic or intravesical chemotherapeutic agent during the study.
* Receiving any other investigational agents.
* The presence of an impaired immune response irrespective of whether this impairment is congenital or caused by disease, drugs or other therapy.
* Known positive HIV serology.
* Presence of a urinary tract infection; treatment should be withheld until urine culture is negative and antibiotic therapy is stopped.
* Trauma to the urinary bladder. In case of gross hematuria, therapy should be stopped or postponed until the hematuria has been successfully treated or has resolved.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BCG vaccine.
* Uncontrolled intercurrent illness.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy: pregnant women are excluded from this study because VERITY-BCG is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with VERITY-BCG, breastfeeding should be discontinued if the mother is treated with VERITY-BCG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) at 24 months | 24 months
  Cumulative Recurrence Free Survival (RFS) at 24 months following 1st intravesical instillation as estimated using the Kaplan - Meier estimator of the survival function.
  Recurrence will be defined as the reappearance of any of the NMIBC tumors as confirmed by cystoscopic biopsy or TURBT.

SECONDARY OUTCOMES:
Recurrence Free Survival (RFS) | 36 months
  Cumulative Recurrence Free Survival (RFS) at 36 months following 1st intravesical instillation as estimated using the Kaplan - Meier estimator of the survival function.
Progression Free Survival (PFS) | 24 months
  Progression Free Survival (PFS) at 24 months as estimated using the Kaplan - Meier estimator of the survival function.
Progression Free Survival (PFS) | 36 months
  Progression Free Survival (PFS) at 36 months as estimated using the Kaplan - Meier estimator of the survival function.
Overall Survival (OS) | 36 months
  Overall Survival (OS) at 36 months as estimated using the Kaplan - Meier estimator of the survival function.
Change in Quality of Life | 36 months
  Change in Quality of Life as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire for NMIBC (EORTC-QLQ-NMIBC24) over 36 months.
  The EORTC QLQ-NMIBC24 is a 24-item self-administered questionnaire that measures health-related quality of life in patients with intermediate to high-risk NMIBC. Items are ranked by the patient from 1 to 4 indicating the extent to which they have experienced those symptoms or problems. 1 = Not at All, 2 = A little, 3=Quite a bit, 4 = Very Much.
  - High Score is equivalent to more problems, except for items on sexual function and sexual enjoyment for which a high score is interpreted as better function.
Change in functioning and symptom status | 36 months
  Change in functioning and symptom status as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire for Cancer Patients (EORTC-QLQ-C30) over 36 months.
  The EORTC QLQ-C30 consists of 30 items and measures Health Related Quality of Life as well as presence of symptoms across all cancer types. The QLQ-C30 includes nine multi-item scales:
  * 5 functional scales (physical, role, cognitive, emotional, and social)
  * 3 symptom scales (fatigue, pain, and nausea and vomiting);
  * A global health and quality-of-life scale*
  * Several single-item symptom measures
    28 Items are ranked 1 to 4. 1 = Not at All, 2 = A little, 3=Quite a bit, 4 = Very Much.
    *2 items are ranked 1 to 7. 1=Very Poor, 7 = Excellent.
  High score = More symptoms or worse problems
  *High Score = Better overall health or Quality of life.

OTHER OUTCOMES:
Safety: Incidence of treatment-emergent AEs and SAEs | 36 months
  Incidence of treatment-emergent AEs and SAEs defined according to the CTCAE v5.0;
Safety: Number of discontinued subjects | 36
  Number of subjects discontinuing study drug due to AEs
Safety: concomitant medications | 36 months
  Usage of concomitant medications over time.

CONTACTS AND LOCATIONS:
Overall Officials: Girish S Kulkarni, MD, Principal Investigator — Princess Margaret Cancer Centre, 700 University Ave, 6-824 Toronto, ON, M5G 1X6, Canada; Alexandre R Zlotta, MD, PhD, FRCSC, Principal Investigator — Mount Sinai Hospital, 600 University Avenue, Toronto, ON, M5G 1X5
Locations (6):
- Canada (6):
  - Site 05, Vancouver, British Columbia
  - Site 04, Kingston, Ontario
  - Site 01, Toronto, Ontario
  - Site 02, Toronto, Ontario
  - Site 08, Toronto, Ontario
  - Site 10, Montreal, Quebec